CLINICAL TRIAL: NCT01636531
Title: A Multi-center, Randomized Open-label, Single-dose, Parallel Group Investigation of the Relative Bioavailability, Tolerability and Dose-exposure Relationship of a High Concentration Liquid Formulation (HCLF) Versus a Lyophilized Formulation (LyoF) of RO4909832 (Gantenerumab) When Administered by su
Brief Title: A Study of A High Concentration Liquid Formulation Versus A Lyophilized Formulation of Gantenerumab in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: WP27951; 2011-006093-65 (EudraCT Number)
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — gantenerumab

ARMS (2):
- HCLF (Experimental)
  Interventions: Drug: gantenerumab
- LyoF (Active Comparator)
  Interventions: Drug: gantenerumab

INTERVENTIONS:
Drug: gantenerumab — High concentration liquid formulation (HCLF), single dose sc
  Arms: HCLF
Drug: gantenerumab — Lyophilized formulation (LyoF), single dose sc
  Arms: LyoF

SUMMARY:
This multi-center, randomized, open-label, single-dose, parallel group study will assess the relative bioavailability, tolerability and dose-exposure relationship of a high concentration liquid formulation (HCLF) versus a lyophilized formulation (LyoF) of gantenerumab (RO4909832) in healthy volunteers. Subjects will be randomized to receive single subcutaneous doses of either HCLF or LyoF. Anticipated time for treatment period and follow-up will be 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 40 to 70 years of age. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history and a complete physical examination
* Body mass index 18.0 to 30.0 kg/m2 inclusive
* Female subjects who are either surgically sterilized or post-menopausal
* Agree not to donate blood or blood products for transfusion for the duration of the study and for one year after their dosing

Exclusion Criteria:

* Suspicion of alcohol or drugs of abuse addiction
* Positive for hepatitis B, hepatitis C or HIV 1 or 2 infection
* Participation in an investigational drug or device study within three months before dosing
* Concomitant disease or condition or treatment which could interfere with the conduct of the study or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Any clinically relevant history of hypersensitivity or allergic reactions, either spontaneous or following drug administration or exposure to food or environmental agents
* Any familial history of early onset Alzheimer's disease
* Claustrophobia, presence of pacemakers, aneurism clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin or body which would contraindicate an MRI scan

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability: Area under the concentration-time curve | Pre-dose and up to 85 days post-dose

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 8 months
Dose-exposure relationship | approximately 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Rennes, France